CLINICAL TRIAL: NCT06143761
Title: A Pilot Study of Neoadjuvant Chemoimmunotherapy in Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Response to Neoadjuvant Chemoimmunotherapy in Resectable Locally Advanced Oral Cancer
Acronym: HNC-SYSU-005
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-184-01
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oral Cancer
Keywords: neoadjuvant chemoimmunotherapy, advanced oral squamous cell carcinoma, therapeutic response, predictive marker, prognosis
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant chemoimmunotherapy+surgery: Patients who underwent neoadjuvant chemoimmunotherapy before surgery
  Interventions: Drug: PD-1 inhibitor+carboplatin+albumin-bound paclitaxel
- surgery: Patients who accepted the surgery alone

INTERVENTIONS:
Drug: PD-1 inhibitor+carboplatin+albumin-bound paclitaxel — A comparative evaluation of patient prognosis between those who received neoadjuvant chemoimmunotherapy-surgery treatment and those who underwent surgery alone.
  Groups: neoadjuvant chemoimmunotherapy+surgery

SUMMARY:
The goal of this observational study is to investigate the effectiveness of neoadjuvant chemoimmunotherapy (NACI) regimens in treating advanced oral squamous cell carcinoma (OSCC) patients. We analyzed clinicopathologic features of advanced OSCC patients who received PD-1 inhibitors in combination with carboplatin and paclitaxel before surgical tumor resection between 2020 and 2022. The Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) and pathologic response were used to evaluate the efficacy of the NACI treatment. Adverse events apparently related to NACI treatment were graded according to the Common Terminology Criteria for Adverse Events, version 4.0. Disease-free survival (DFS) and overall survival (OS) were calculated using the Kaplan-Meier survival curves and compared using the log rank test. Additionally, we calculated the area under curve (AUC) to compare the predictive value of PD-L1 expression with baseline serum lipid biomarkers for patient response.

ELIGIBILITY:
Inclusion Criteria:

Patients with advanced OSCC who received NACI before surgery

* Confirmation of primary OSCC by two experienced pathologists;
* Clinical stage III/ IVA (cT1-2/cN1-2/M0 or cT3-4a/cN0-2/M0) according to the 8th Edition of American Joint Committee on Cancer (AJCC) guideline;
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* No prior anti-cancer therapy;
* Locally resectable advanced tumor evaluated by a head and neck surgeon.

Advanced OSCC patients who only received surgery

* A histopathologic diagnosis of primary OSCC;
* A clinical stage of III/IVA (AJCC, 8th edition);
* An ECOG performance status of 0 to 1.

Exclusion Criteria:

Patients with advanced OSCC who received NACI before surgery

* Patients with other pathological types, without NACI or Surgery;
* Incomplete pre-treatment data;
* Lost to follow up were excluded from the study.

Advanced OSCC patients who only received surgery

* Patients who had received other therapies targeting the head and neck region before the surgery or those with evidence of recurrence or metastasis, as assessed by physical examination reports or imaging studies before surgery
* Lost to follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients underwent NACI before surgery
  * Patients accepted the surgery alone.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  The time(years) from day 1 of study treatment until death from any cause.
Disease-free survival （DFS） | 2 years
  DFS(by months) is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease DFS is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Li, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided